CLINICAL TRIAL: NCT04244760
Title: Peri-operative Pain Assessment in Children Undergoing Orthopaedic Surgery
Brief Title: Pain Assessment in Children Undergoing Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catherine Ferland (Other)
Responsible Party: Sponsor-Investigator, Catherine Ferland, Clinical Researcher, Shriners Hospitals for Children
Organization: Shriners Hospitals for Children (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A08M7114B
Record Dates: First submitted 2020-01-10; First posted 2020-01-28 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Adolescent Idiopathic Scoliosis; Cerebral Palsy
Keywords: Adolescent Idiopathic Scoliosis; Cerebral Palsy; Conditioned Pain Modulation; Chronic Postsurgical Pain; Quantitative Sensory Testing; Pain Management
MeSH Terms: conditions — Cerebral Palsy; Pain, Postoperative; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verbal Patients (Active Comparator)
  Interventions: Behavioral: Pain assessment for verbal patients
- Non-verbal Patients (Active Comparator)
  Interventions: Behavioral: Pain assessment for non-verbal patients

INTERVENTIONS:
Behavioral: Pain assessment for verbal patients — The pain profile of the patient will be assessed at each time point including biological sample analysis (blood and saliva), quantitative sensory testing (mechanical and thermal), and psychological state via the completion of questionnaires by the patient.
  Arms: Verbal Patients
Behavioral: Pain assessment for non-verbal patients — The pain profile of the patient will be assessed at each time point including biological sample analysis (blood and saliva), quantitative sensory testing (mechanical), and psychological state via the completion of questionnaires by the parent of the patient.
  Arms: Non-verbal Patients

SUMMARY:
Musculoskeletal (MSK) pain is one of the most common types of pain among children and adolescents. Recurring episodes of MSK pain conditions have a major impact on the daily lives. Children and adolescents with neuromuscular diseases are often unable to report the pain the patients experience because of intellectual and/or physical limitations. There is no reason to believe that pain is any less frequent or intense in these patients than in normally developing patients. Because of the elusive nature of pain in non-verbal children, therapeutic decisions are frequently based on vague proxy measures of pain and revert to a series of trials and errors. This project creates a unique opportunity to directly characterize and compare MSK and surgical pain subjectively in two different patient samples (verbal and non-verbal). The ultimate goal is to use this information to offer the highest quality of pain control in children with MSK conditions, and more specifically in children with limited communication skills unable to communicate their distress associated with the surgical procedural.

DETAILED DESCRIPTION:
Improvement in the assessment techniques, to enable better pain management in children with intellectual and developmental disabilities who are unable to describe the intensity of the postsurgical pain, is a cornerstone of our research program. This research project will elucidate the regulation of specific markers of global surgical insult (nociception, inflammation, stress responses) associated to specific physiological mechanisms related to pain in children with and without verbal skills undergoing major orthopaedic surgery. This project creates a unique opportunity to directly characterize and compare MSK and surgical pain subjectively in the two different patient samples (verbal and non-verbal). As molecular events of pathophysiological processes are quantifiable, the investigators will test for associations between the expression of front-running pain biomarkers in physiological fluids (blood and saliva) and the experience of pain in two patient samples (verbal and non-verbal) undergoing major orthopaedic surgery. The identification of biomarkers will provide a deeper understanding of a patient's pain perception alongside self-report or observers' report subjective measurements. Even with standardization of best practice perioperative anesthetic pain management, children undergoing similar surgical procedures experience pain at different intensity. Based on preliminary findings, treatment modalities appear to be ineffective in one out of five patients. Pain experience variability may originate in the lack of rigor in the clinical pain assessment tools. Tools such as numerical rating scales used in the perioperative period are not based on objective patient specific pain thresholds. A personalized mechanism-based approach may be the key to better identify a patient's postsurgical pain outcome and how this assessment could lead to personalized perioperative pain management. The ultimate goal is to use this information to offer the highest quality of pain control in children with MSK conditions, and more specifically in children with limited communication skills unable to communicate their distress associated with the surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 10 and 21 years old
* Scheduled to undergo posterior or anterior spinal fusion surgery for AIS with instrumentation
* Ability to adequately understand and respond to outcome measures
* No previous major orthopedic surgery
* Female or male
* Any ethnic background

Exclusion Criteria:

* Inability of the child to speak English or French
* Diagnosed with developmental delay that would interfere with understanding questions being asked (autism, mental retardation)
* Children with major chronic medical conditions (ASA status III or higher)

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Pain intensity as assessed by the The Faces Pain Scale -Revised (0-10 scale, with higher score indicating more pain) in verbal patients | Baseline
Pain intensity as assessed by the The Faces Pain Scale -Revised (0-10 scale, with higher score indicating more pain) in verbal patients | Postoperative day 1
Pain intensity as assessed by the The Faces Pain Scale -Revised (0-10 scale, with higher score indicating more pain) in verbal patients | Postoperative day 2
Pain intensity as assessed by the The Faces Pain Scale -Revised (0-10 scale, with higher score indicating more pain) in verbal patients | Postoperative day 5
Pain intensity as assessed by the The Faces Pain Scale -Revised (0-10 scale, with higher score indicating more pain) in verbal patients | 6 weeks postoperative
Pain intensity as assessed by the The Faces Pain Scale -Revised (0-10 scale, with higher score indicating more pain) in verbal patients | 6 months postoperative
Pain intensity as assessed by the The Faces Pain Scale -Revised (0-10 scale, with higher score indicating more pain) in verbal patients | 1 year postoperative
Pain intensity as assessed by the The Faces Pain Scale -Revised (0-10 scale, with higher score indicating more pain) in verbal patients | 2 years postoperative
Pain intensity as assessed by the Non-Communicating Children's Pain Checklist-Revised (NCCPC-R), and its post-operative version in non-verbal patients, with higher score indicating more pain | Baseline
Pain intensity as assessed by the Non-Communicating Children's Pain Checklist-Revised (NCCPC-R), and its post-operative version in non-verbal patients, with higher score indicating more pain | Postoperative day 1
Pain intensity as assessed by the Non-Communicating Children's Pain Checklist-Revised (NCCPC-R), and its post-operative version in non-verbal patients, with higher score indicating more pain | Postoperative day 2
Pain intensity as assessed by the Non-Communicating Children's Pain Checklist-Revised (NCCPC-R), and its post-operative version in non-verbal patients, with higher score indicating more pain | Postoperative day 5
Pain intensity as assessed by the Non-Communicating Children's Pain Checklist-Revised (NCCPC-R), and its post-operative version in non-verbal patients, with higher score indicating more pain | 6 weeks postoperative
Pain intensity as assessed by the Non-Communicating Children's Pain Checklist-Revised (NCCPC-R), and its post-operative version in non-verbal patients, with higher score indicating more pain | 6 months postoperative
Pain intensity as assessed by the Non-Communicating Children's Pain Checklist-Revised (NCCPC-R), and its post-operative version in non-verbal patients, with higher score indicating more pain | 1 year postoperative
Pain intensity as assessed by the Non-Communicating Children's Pain Checklist-Revised (NCCPC-R), and its post-operative version in non-verbal patients, with higher score indicating more pain | 2 years postoperative

SECONDARY OUTCOMES:
Mechanical detection threshold (grams) as measured with von Frey filaments | Baseline
Pain pressure threshold (Newtons) as measured with an algometer. | Baseline
Conditioned pain modulation (CPM) efficiency, a physiological parameter calculated as the percentage difference between the average pain intensity (0-10) reported during a thermode (heat) test before and after a cold water submersion bath test. | Baseline
  Conditioned pain modulation measurement is omitted in the non-verbal patient arm.
Mechanical detection threshold (grams) as measured with von Frey filaments | Postoperative day 1
Pain pressure threshold (Newtons) as measured with an algometer. | Postoperative day 1
Mechanical detection threshold (grams) as measured with von Frey filaments | Postoperative day 2
Pain pressure threshold (Newtons) as measured with an algometer. | Postoperative day 2
Mechanical detection threshold (grams) as measured with von Frey filaments | Postoperative day 5
Pain pressure threshold (Newtons) as measured with an algometer. | Postoperative day 5
Conditioned pain modulation (CPM) efficiency, a physiological parameter calculated as the percentage difference between the average pain intensity (0-10) reported during a thermode (heat) test before and after a cold water submersion bath test. | Postoperative day 5
  Conditioned pain modulation measurement is omitted in the non-verbal patient arm.
Mechanical detection threshold (grams) as measured with von Frey filaments | 6 weeks postoperative
Pain pressure threshold (Newtons) as measured with an algometer. | 6 weeks postoperative
Conditioned pain modulation (CPM) efficiency, a physiological parameter calculated as the percentage difference between the average pain intensity (0-10) reported during a thermode (heat) test before and after a cold water submersion bath test. | 6 weeks postoperative
  Conditioned pain modulation measurement is omitted in the non-verbal patient arm.
Mechanical detection threshold (grams) as measured with von Frey filaments | 6 months postoperative
Pain pressure threshold (Newtons) as measured with an algometer. | 6 months postoperative
Conditioned pain modulation (CPM) efficiency, a physiological parameter calculated as the percentage difference between the average pain intensity (0-10) reported during a thermode (heat) test before and after a cold water submersion bath test. | 6 months postoperative
  Conditioned pain modulation measurement is omitted in the non-verbal patient arm.
Mechanical detection threshold (grams) as measured with von Frey filaments | 1 year postoperative
Pain pressure threshold (Newtons) as measured with an algometer. | 1 year postoperative
Conditioned pain modulation (CPM) efficiency, a physiological parameter calculated as the percentage difference between the average pain intensity (0-10) reported during a thermode (heat) test before and after a cold water submersion bath test. | 1 year postoperative
  Conditioned pain modulation measurement is omitted in the non-verbal patient arm.
Mechanical detection threshold (grams) as measured with von Frey filaments | 2 years postoperative
Pain pressure threshold (Newtons) as measured with an algometer. | 2 years postoperative
Conditioned pain modulation (CPM) efficiency, a physiological parameter calculated as the percentage difference between the average pain intensity (0-10) reported during a thermode (heat) test before and after a cold water submersion bath test. | 2 years postoperative
  Conditioned pain modulation measurement is omitted in the non-verbal patient arm.
Total Score of the Pain Catastrophizing Scale (0-52). Higher scores indicate higher levels of pain-related anxiety. | Baseline
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Total Score of the Pain Catastrophizing Scale (0-52). Higher scores indicate higher levels of pain-related anxiety. | Postoperative day 1
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Total Score of the Pain Catastrophizing Scale (0-52). Higher scores indicate higher levels of pain-related anxiety. | Postoperative day 2
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Total Score of the Pain Catastrophizing Scale (0-52). Higher scores indicate higher levels of pain-related anxiety. | Postoperative day 5
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Total Score of the Pain Catastrophizing Scale (0-52). Higher scores indicate higher levels of pain-related anxiety. | 6 weeks postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Total Score of the Pain Catastrophizing Scale (0-52). Higher scores indicate higher levels of pain-related anxiety. | 6 months postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Total Score of the Pain Catastrophizing Scale (0-52). Higher scores indicate higher levels of pain-related anxiety. | 1 year postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Total Score of the Pain Catastrophizing Scale (0-52). Higher scores indicate higher levels of pain-related anxiety. | 2 years postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Total score (30-150) across to 4 domains of the Scoliosis Research Society Questionnaire-30 (SRS-30) regarding the outcome of the patient's spine surgery (items scored from 1=worst, to 5=best, thus lower scores mean worse outcomes). | Baseline
  4 domains: 1) pain (max. score 30) 2) mental health (max. score 25) 3) function/activity (max. score 35) 4) Self Image/appearance (max. score 45)
Total score (30-150) across to 4 domains of the Scoliosis Research Society Questionnaire-30 (SRS-30) regarding the outcome of the patient's spine surgery (items scored from 1=worst, to 5=best, thus lower scores mean worse outcomes). | 6 weeks postoperative
  4 domains: 1) pain (max. score 30) 2) mental health (max. score 25) 3) function/activity (max. score 35) 4) Self Image/appearance (max. score 45)
Total score (30-150) across to 4 domains of the Scoliosis Research Society Questionnaire-30 (SRS-30) regarding the outcome of the patient's spine surgery (items scored from 1=worst, to 5=best, thus lower scores mean worse outcomes). | 6 months postoperative
  4 domains: 1) pain (max. score 30) 2) mental health (max. score 25) 3) function/activity (max. score 35) 4) Self Image/appearance (max. score 45)
Total score (30-150) across to 4 domains of the Scoliosis Research Society Questionnaire-30 (SRS-30) regarding the outcome of the patient's spine surgery (items scored from 1=worst, to 5=best, thus lower scores mean worse outcomes). | 1 year postoperative
  4 domains: 1) pain (max. score 30) 2) mental health (max. score 25) 3) function/activity (max. score 35) 4) Self Image/appearance (max. score 45)
Total score (30-150) across to 4 domains of the Scoliosis Research Society Questionnaire-30 (SRS-30) regarding the outcome of the patient's spine surgery (items scored from 1=worst, to 5=best, thus lower scores mean worse outcomes). | 2 years postoperative
  4 domains: 1) pain (max. score 30) 2) mental health (max. score 25) 3) function/activity (max. score 35) 4) Self Image/appearance (max. score 45)
Total Score of the Functional Disability Inquiry (0-60). Higher scores indicate greater activity limitations during the past 2 weeks. | Baseline
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Total Score of the Functional Disability Inquiry (0-60). Higher scores indicate greater activity limitations during the past 2 weeks. | 6 weeks postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Total Score of the Functional Disability Inquiry (0-60). Higher scores indicate greater activity limitations during the past 2 weeks. | 6 months postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Total Score of the Functional Disability Inquiry (0-60). Higher scores indicate greater activity limitations during the past 2 weeks. | 1 year postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Total Score of the Functional Disability Inquiry (0-60). Higher scores indicate greater activity limitations during the past 2 weeks. | 2 years postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Score of State Anxiety of the State-Trait Anxiety Scale (20-60). Higher scores indicate greater state anxiety. | Baseline
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Score of Trait Anxiety of the State-Trait Anxiety Scale (20-60). Higher scores indicate greater trait anxiety. | Baseline
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Score of State Anxiety of the State-Trait Anxiety Scale (20-60). Higher scores indicate greater state anxiety. | Day of surgery
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Score of Trait Anxiety of the State-Trait Anxiety Scale (20-60). Higher scores indicate greater trait anxiety. | Day of surgery
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Score of State Anxiety of the State-Trait Anxiety Scale (20-60). Higher scores indicate greater state anxiety. | 6 weeks postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Score of Trait Anxiety of the State-Trait Anxiety Scale (20-60). Higher scores indicate greater trait anxiety. | 6 weeks postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Score of State Anxiety of the State-Trait Anxiety Scale (20-60). Higher scores indicate greater state anxiety. | 6 months postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Score of Trait Anxiety of the State-Trait Anxiety Scale (20-60). Higher scores indicate greater trait anxiety. | 6 months postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Score of State Anxiety of the State-Trait Anxiety Scale (20-60). Higher scores indicate greater state anxiety. | 1 year postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Score of Trait Anxiety of the State-Trait Anxiety Scale (20-60). Higher scores indicate greater trait anxiety. | 1 year postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Score of State Anxiety of the State-Trait Anxiety Scale (20-60). Higher scores indicate greater state anxiety. | 2 years postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Score of Trait Anxiety of the State-Trait Anxiety Scale (20-60). Higher scores indicate greater trait anxiety. | 2 years postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Score on Activity Avoidance and Somatic Function of the Tampa Scale for Kinesiophobia (score 17-68). Higher scores indicate greater kinesiophobia. | Baseline
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Score on Activity Avoidance and Somatic Function of the Tampa Scale for Kinesiophobia (score 17-68). Higher scores indicate greater kinesiophobia. | Postoperative day 1
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Score on Activity Avoidance and Somatic Function of the Tampa Scale for Kinesiophobia (score 17-68). Higher scores indicate greater kinesiophobia. | Postoperative day 2
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Score on Activity Avoidance and Somatic Function of the Tampa Scale for Kinesiophobia (score 17-68). Higher scores indicate greater kinesiophobia. | Postoperative day 5
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Score on Activity Avoidance and Somatic Function of the Tampa Scale for Kinesiophobia (score 17-68). Higher scores indicate greater kinesiophobia. | 6 weeks postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Score on Activity Avoidance and Somatic Function of the Tampa Scale for Kinesiophobia (score 17-68). Higher scores indicate greater kinesiophobia. | 6 months postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Score on Activity Avoidance and Somatic Function of the Tampa Scale for Kinesiophobia (score 17-68). Higher scores indicate greater kinesiophobia. | 1 year postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Score on Activity Avoidance and Somatic Function of the Tampa Scale for Kinesiophobia (score 17-68). Higher scores indicate greater kinesiophobia. | 2 years postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Global Score of the Pittsburgh Sleep Quality Index (0-21). Higher scores indicate a worse sleep quality (>5 indicates "poor sleeper"). | Baseline
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Global Score of the Pittsburgh Sleep Quality Index (0-21). Higher scores indicate a worse sleep quality (>5 indicates "poor sleeper"). | Postoperative day 1
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Global Score of the Pittsburgh Sleep Quality Index (0-21). Higher scores indicate a worse sleep quality (>5 indicates "poor sleeper"). | Postoperative day 2
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Global Score of the Pittsburgh Sleep Quality Index (0-21). Higher scores indicate a worse sleep quality (>5 indicates "poor sleeper"). | Postoperative day 5
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Global Score of the Pittsburgh Sleep Quality Index (0-21). Higher scores indicate a worse sleep quality (>5 indicates "poor sleeper"). | 6 weeks postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Global Score of the Pittsburgh Sleep Quality Index (0-21). Higher scores indicate a worse sleep quality (>5 indicates "poor sleeper"). | 6 months postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Global Score of the Pittsburgh Sleep Quality Index (0-21). Higher scores indicate a worse sleep quality (>5 indicates "poor sleeper"). | 1 year postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.
Global Score of the Pittsburgh Sleep Quality Index (0-21). Higher scores indicate a worse sleep quality (>5 indicates "poor sleeper"). | 2 years postoperative
  Completed by patient in verbal patient arm and by parent of the patient in non-verbal patient arm.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Ferland, Principal Investigator — Shriners Hospitals for Children,Canada
Locations (1):
- Shriners Hospital for Children-Canada, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No